CLINICAL TRIAL: NCT07040293
Title: Evaluation of the Efficacy and Safety of Absorbable Bone Wax and Traditional Bone Wax for Facet Fusion After Lumbar Fusion Surgery: A Multicenter, Randomized, Open-label, Superiority Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Absorbable vs Traditional Bone Wax for Facet Fusion After Lumbar Fusion Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Jiangxi Provincial People's Hopital (Other); The First Affiliated Hospital of Nanchang University (Other); Qilu Hospital of Shandong University (Other); Beijing Chao Yang Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Principal Investigator, Haifeng Wei, MD, PhD, vice director, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024SL158
Record Dates: First submitted 2025-06-15; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Fusion Surgery; Fusion of Joint
Keywords: absorbable bone wax; traditional bone wax; facet fusion after lumbar fusion surgery; hemostasis
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absorbable bone wax gruop (Experimental)
  Interventions: Device: Absorbable bone wax for hemostasis in the osteotomy surface of the facet joint
- Traditional bone wax group (Active Comparator)
  Interventions: Device: Traditional bone wax for hemostasis in the osteotomy surface of the facet joint

INTERVENTIONS:
Device: Absorbable bone wax for hemostasis in the osteotomy surface of the facet joint — Following the enrollment of patients who underwent posterior lumbar decompression, intervertebral bone graft, and internal fixation surgery, a "V-shaped" osteotomy was executed at the facet joint contralateral to the decompression site, with 0.5g absorbable bone wax subsequently applied to the osteotomy surface.
  Arms: Absorbable bone wax gruop
Device: Traditional bone wax for hemostasis in the osteotomy surface of the facet joint — Following the enrollment of patients who underwent posterior lumbar decompression, intervertebral bone graft fusion, and internal fixation surgery, a "V-shaped" osteotomy was executed at the facet joint contralateral to the decompression site, with 0.5g traditional bone wax subsequently applied to the osteotomy surface.
  Arms: Traditional bone wax group

SUMMARY:
Hemorrhage on the surface of cancellous bone presents a significant challenge in orthopedic surgery. Traditional bone wax, commonly utilized for hemostasis in bone wounds, is non-absorbable and associated with various complications, including pseudarthrosis, paralysis, venous sinus thrombosis, chronic inflammation, allergic reactions, and infections, thereby limiting its clinical utility. In contrast, absorbable bone wax, primarily composed of medical-grade water-soluble polymer materials, exhibits excellent biocompatibility. It is fully absorbed, excreted, or eliminated by the body without leaving toxic residues. This study employs a rigorous efficacy design to select an appropriate patient cohort for lumbar fusion surgery, based on specific inclusion and exclusion criteria. Participants are randomly assigned to either an experimental group receiving absorbable bone wax or a control group receiving traditional bone wax, facilitating a randomized, open-label, parallel-controlled clinical trial. This study aims to evaluate the comparative effects of absorbable bone wax versus traditional bone wax on the rate of bone fusion following hemostasis of bone wounds. The objective is to furnish robust evidence-based insights into the application of absorbable bone wax for bone wounds necessitating fusion, thereby establishing a safe, effective, and broadly applicable technique for bone wound hemostasis in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged between 18 and 75 years, with no restrictions on gender.
* Participants with conditions such as single-segment lumbar intervertebral disc protrusion, lumbar spondylolisthesis, and lumbar spinal stenosis who are scheduled to undergo posterior decompression, intervertebral fusion, and internal fixation surgery.
* Participants must be able to comprehend the objectives of the study, willingly participate, and provide informed consent by signing the consent form.

Exclusion Criteria:

* Individuals with a hemorrhagic predisposition or coagulation disorders, indicated by a prothrombin time (PT) of 18 seconds or greater, and those with a history of prolonged anticoagulant use.
* Individuals presenting with lumbar spine infections or fractures.
* Individuals with known allergies to materials such as polyethylene glycol, sodium carboxymethyl cellulose, and bone wax (including beeswax, paraffin, and isopropyl palmitate).
* Individuals whose conditions are critical, making it challenging to accurately assess the efficacy and safety of the equipment.
* Individuals deemed by researchers to have poor compliance, rendering them unable to fulfill the study requirements.
* Women who are currently pregnant, intend to become pregnant within the past year, or are breastfeeding.
* Individuals who have participated in other clinical trials within the preceding 30 days to prevent cross-interference.
* Individuals with significant complications or comorbidities, such as severe cardiovascular, hepatic, renal, or other chronic conditions that could influence surgical risks and research outcomes.
* Individuals identified by researchers as having a life expectancy of less than six months.
* Individuals with severe osteoporosis, defined as a bone mineral density T-score of ≤-2.5 accompanied by fragility fractures.
* Any other individuals deemed unsuitable for participation in this clinical trial by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The clinical fusion rate of lumbar facet joints | 6 months
  The proportion of individuals achieving the clinical fusion standard of the facet joint was assessed within each group. Six months postoperatively, the fusion status of the facet joints at the surgical segments was evaluated using continuous thin-slice CT plain scans combined with three-dimensional reconstruction images of the lumbar vertebrae. The evaluation criteria were based on the guidelines established by Ren et al. (2020) in their study on modified facet joint fusion for lumbar degenerative disease. According to these criteria, clinical fusion is confirmed when one side of the facet joint attains grade I or grade II radiological fusion standards.

SECONDARY OUTCOMES:
The success rate of hemostasis within three minutes | 3 minutes
  The success rate of achieving hemostasis within three minutes during surgery is defined as the proportion of patients who meet the hemostatic objective within this timeframe.
Postoperative wound healing | 14 days
  Postoperative wound healing is assessed 14 days following the procedure, with observations including the presence of bleeding, redness, and swelling at the wound site.

OTHER OUTCOMES:
Incidence of adverse events | 6 months
  This encompasses any adverse events associated with the use of bone wax, such as infections, inflammatory responses, and allergic reactions.
Postoperative infection rate | 6 months
  This metric evaluates the frequency of infections occurring in the surgical area and serves as a critical indicator of surgical safety.
Reoperation rate | 6 months
  This refers to the proportion of cases requiring additional surgical intervention due to unsuccessful hemostasis or other complications.
Long-term complications | 6 months
  This includes any complications or adverse reactions related to the use of bone wax that manifest during the extended postoperative follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ren Z, Li Z, Li S, Xu D, Chen X. Modified Facet Joint Fusion for Lumbar Degenerative Disease: Case Series of a Fusion Technique, Clinical Outcomes, and Fusion Rate in 491 Patients. Oper Neurosurg. 2020 Sep 1;19(3):255-263. doi: 10.1093/ons/opaa147. PMID 32469075
- [Background] Vestergaard RF, Nielsen PH, Terp KA, Soballe K, Andersen G, Hasenkam JM. Effect of hemostatic material on sternal healing after cardiac surgery. Ann Thorac Surg. 2014 Jan;97(1):153-60. doi: 10.1016/j.athoracsur.2013.08.030. Epub 2013 Oct 8. PMID 24119983
- [Background] An KC, Kong GM, Park DH, Baik JM, Youn JH, Lee WS. Comparison of Posterior Lumbar Interbody Fusion and Posterolateral Lumbar Fusion in Monosegmental Vacuum Phenomenon within an Intervertebral Disc. Asian Spine J. 2016 Feb;10(1):93-8. doi: 10.4184/asj.2016.10.1.93. Epub 2016 Feb 16. PMID 26949464
- [Background] Kim JG, Ham DW, Zheng H, Kwon O, Kim HJ. Evaluating the Efficacy of Water-Soluble Bone Wax (Tableau Wax) in Reducing Blood Loss in Spinal Fusion Surgery: A Randomized, Controlled, Pilot Study. Medicina (Kaunas). 2023 Aug 25;59(9):1545. doi: 10.3390/medicina59091545. PMID 37763664
- [Background] Wang R, Jin Z, Gao J, Ma Y, Han Q. Effectiveness and Biocompatibility Evaluation of a Novel Absorbable Bone Wax Used in Bone Tissue. Tissue Eng Part C Methods. 2024 Aug;30(8):353-363. doi: 10.1089/ten.TEC.2024.0144. PMID 39113538
- [Background] Duan Q, Liu H, Zheng L, Cai D, Huang G, Liu Y, Guo R. Novel resorbable bone wax containing beta-TCP and starch microspheres for accelerating bone hemostasis and promoting regeneration. Front Bioeng Biotechnol. 2023 Jan 19;11:1105306. doi: 10.3389/fbioe.2023.1105306. eCollection 2023. PMID 36741749
- [Background] Choi SY, Rhim J, Heo SA, Han WJ, Kim MH, Ha CW. Efficacy and safety of a novel hemostatic material, BoneStat, compared with Ostene and Bone Wax in a rat calvarial defect model. Int J Artif Organs. 2021 Oct;44(10):734-747. doi: 10.1177/03913988211021428. Epub 2021 Aug 13. PMID 34387533
- [Background] Tham T, Roberts K, Shanahan J, Burban J, Costantino P. Analysis of bone healing with a novel bone wax substitute compared with bone wax in a porcine bone defect model. Future Sci OA. 2018 Jul 26;4(8):FSO326. doi: 10.4155/fsoa-2018-0004. eCollection 2018 Sep. PMID 30271614
- [Background] Wellisz T, An YH, Wen X, Kang Q, Hill CM, Armstrong JK. Infection rates and healing using bone wax and a soluble polymer material. Clin Orthop Relat Res. 2008 Feb;466(2):481-6. doi: 10.1007/s11999-007-0067-5. Epub 2008 Jan 10. PMID 18196435
- [Background] Gibbs L, Kakis A, Weinstein P, Conte JE Jr. Bone wax as a risk factor for surgical-site infection following neurospinal surgery. Infect Control Hosp Epidemiol. 2004 Apr;25(4):346-8. doi: 10.1086/502403. PMID 15108734
- [Background] Schonauer C, Tessitore E, Barbagallo G, Albanese V, Moraci A. The use of local agents: bone wax, gelatin, collagen, oxidized cellulose. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S89-96. doi: 10.1007/s00586-004-0727-z. Epub 2004 Jun 22. PMID 15221572
- [Background] Julsrud ME. A surgical complication: allergic reaction to bone wax. J Foot Surg. 1980 Fall;19(3):152-4. No abstract available. PMID 7021652
- [Background] Solomon LB, Guevara C, Buchler L, Howie DW, Byard RW, Beck M. Does bone wax induce a chronic inflammatory articular reaction? Clin Orthop Relat Res. 2012 Nov;470(11):3207-12. doi: 10.1007/s11999-012-2457-6. Epub 2012 Jul 4. PMID 22760602
- [Background] Crocker M, Nesbitt A, Rich P, Bell B. Symptomatic venous sinus thrombosis following bone wax application to emissary veins. Br J Neurosurg. 2008 Dec;22(6):798-800. doi: 10.1080/02688690802256399. PMID 19085366
- [Background] Stein JM, Eskey CJ, Mamourian AC. Mass effect in the thoracic spine from remnant bone wax: an MR imaging pitfall. AJNR Am J Neuroradiol. 2010 May;31(5):844-6. doi: 10.3174/ajnr.A1830. Epub 2009 Nov 12. PMID 19910449
- [Background] Kumar A, Kale SS, Dutta R, Kumar A. Post-thoracotomy paraplegia due to epidural migration of bone wax. Eur J Cardiothorac Surg. 2009 Apr;35(4):734-6. doi: 10.1016/j.ejcts.2008.11.037. Epub 2009 Feb 23. PMID 19233676
- [Background] Angelini GD, el-Ghamari FA, Butchart EG. Poststernotomy pseudo-arthrosis due to foreign body reaction to bone wax. Eur J Cardiothorac Surg. 1987;1(2):129-30. doi: 10.1016/1010-7940(87)90025-x. PMID 2856608